CLINICAL TRIAL: NCT05514327
Title: the Safety and Efficacy of Ultra-fraction Radiotherapy Bridging CART Cell Therapy in Relapsed/Refractory Diffuse Large b Cell Lymphoma
Brief Title: A Study of Ultra-fraction Radiotherapy Bridging CART in R/R DLBCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Ruanjing, Docter, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART-1
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Diffuse Large B Cell Lymphoma; CAR-T; Radiotherapy; Bridging Therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): ultra-fraction radiotherapy + CAR-T
  Interventions: Radiation: ultra-fraction radiotherapy

INTERVENTIONS:
Radiation: ultra-fraction radiotherapy — the R/R DLBCL patients would receive ultra-fraction radiotherapy as bridging therapy before the CD19 CART cell infusion

SUMMARY:
This is a single-arm single center study to prospectively evaluate the safety and efficacy of ultra-fraction radiotherapy bridging CAR-T therapy in relapsed/refractory diffuse large b cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Over than 18 years old
2. Histologically confirmed DLBCL(by central pathology review before enrolment)
3. Relapsed or refractory disease after ≥2 lines of chemotherapy including rituximab and anthracycline and either having failed autologous Hematopoietic stem cell transplantation (ASCT), or being ineligible for or not consenting to ASCT
4. Measurable disease at time of enrollment (the maximum diameter of cross section ≥1.5cm)
5. Life expectancy ≥12 weeks
6. Able to receive radiotherapy evaluated by specialist

Exclusion Criteria:

1. Prior radiation therapy within 1 year of infusion
2. Pregnant or nursing (lactating) women
3. Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
4. Previous solid tumor within 3 years, previous or concurrent hematological malignancy
5. Severe organ dysfunction: left ventricle ejection fraction (LVEF) <40%; DLCO <40%; estimated glomerular filtration rate (eGFR)<30mL/min/1.73 m2; total bilirubin >3 ULN
6. HIV positive patients, active replication of or prior infection with hepatitis B or active hepatitis C( HCV RNA positive );
7. Other conditions that the investigator may exclude due to risks or other possibilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
3-month ORR | 3 months
  the overall response rate at 3 months after CAR-T cell infusion

SECONDARY OUTCOMES:
2-year PFS | 2 years
  the 2-year progression free survival time from CAR-T cell infusion
2-year OS | 2 years
  the 2-year overall survival time from CAR-T cell infusion
6-month ORR | 6 months
  the overall response rate at 6 months after CAR-T cell infusion
DOR | 2 years
  the duration of response time
relapse rate | 2 years
  the cumulative rate of relapse
the rate of severe side effects | 2 years
  the rate of severe side effects (CTCAE≥ grade 3）

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
the study protocol, statistical analysis plan, informed consent form, clinical study report would be available upon email request in 3 years after the closure of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years after the closure of the study
Access Criteria: upon email request

REFERENCES:
- [Background] Minn I, Rowe SP, Pomper MG. Enhancing CAR T-cell therapy through cellular imaging and radiotherapy. Lancet Oncol. 2019 Aug;20(8):e443-e451. doi: 10.1016/S1470-2045(19)30461-9. Epub 2019 Jul 29. PMID 31364596
- [Background] Kuhnl A, Roddie C, Kirkwood AA, Tholouli E, Menne T, Patel A, Besley C, Chaganti S, Sanderson R, O'Reilly M, Norman J, Osborne W, Bloor A, Lugthart S, Malladi R, Patten PEM, Neill L, Martinez-Cibrian N, Kennedy H, Phillips EH, Jones C, Sharplin K, El-Sharkawi D, Latif AL, Mathew A, Uttenthal B, Stewart O, Marzolini MAV, Townsend W, Cwynarski K, Ardeshna K, Ardavan A, Robinson K, Pagliuca A, Collins GP, Johnson R, McMillan A. A national service for delivering CD19 CAR-Tin large B-cell lymphoma - The UK real-world experience. Br J Haematol. 2022 Aug;198(3):492-502. doi: 10.1111/bjh.18209. Epub 2022 Apr 29. PMID 35485402
- [Background] Qu C, Ping N, Kang L, Liu H, Qin S, Wu Q, Chen X, Zhou M, Xia F, Ye A, Kong D, Li C, Yu L, Wu D, Jin Z. Radiation Priming Chimeric Antigen Receptor T-Cell Therapy in Relapsed/Refractory Diffuse Large B-Cell Lymphoma With High Tumor Burden. J Immunother. 2020 Jan;43(1):32-37. doi: 10.1097/CJI.0000000000000284. PMID 31219975
- [Background] Sim AJ, Jain MD, Figura NB, Chavez JC, Shah BD, Khimani F, Lazaryan A, Krivenko G, Davila ML, Liu HD, Falchook AD, Dahiya S, Rapoport AP, Kim S, Locke FL, Robinson TJ. Radiation Therapy as a Bridging Strategy for CAR T Cell Therapy With Axicabtagene Ciloleucel in Diffuse Large B-Cell Lymphoma. Int J Radiat Oncol Biol Phys. 2019 Dec 1;105(5):1012-1021. doi: 10.1016/j.ijrobp.2019.05.065. Epub 2019 Jun 5. PMID 31175906
- [Background] Manjunath SH, Cohen AD, Lacey SF, Davis MM, Garfall AL, Melenhorst JJ, Maxwell R, Arscott WT, Maity A, Jones JA, Plastaras JP, Stadtmauer EA, Levine BL, June CH, Milone MC, Paydar I. The Safety of Bridging Radiation with Anti-BCMA CAR T-Cell Therapy for Multiple Myeloma. Clin Cancer Res. 2021 Dec 1;27(23):6580-6590. doi: 10.1158/1078-0432.CCR-21-0308. Epub 2021 Sep 15. PMID 34526365
- [Background] DeSelm C, Palomba ML, Yahalom J, Hamieh M, Eyquem J, Rajasekhar VK, Sadelain M. Low-Dose Radiation Conditioning Enables CAR T Cells to Mitigate Antigen Escape. Mol Ther. 2018 Nov 7;26(11):2542-2552. doi: 10.1016/j.ymthe.2018.09.008. Epub 2018 Sep 13. PMID 30415658